CLINICAL TRIAL: NCT02677844
Title: A Randomized, Single-Blind, Placebo-Controlled, Single Ascending Dose Study to Determine the Exposure-Response Relationship Between Abemaciclib and QT Interval in Healthy Subjects
Brief Title: A Study of Abemaciclib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 16080; I3Y-MC-JPCA (Other: Eli Lilly and Company)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-12

CONDITIONS: Healthy
MeSH Terms: interventions — abemaciclib; Loperamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Abemaciclib (Experimental): 200 - 600 mg single increasing oral dose of abemaciclib on Day 1 of up to 3 study periods.
  Interventions: Drug: Abemaciclib
- Placebo (Placebo Comparator): Single oral dose of placebo on Day 1 of 1 study period.
  Interventions: Drug: Placebo
- Loperamide (Active Comparator): Cohort 2, only. 8 mg Loperamide given orally once in 1 of 4 study periods.
  Interventions: Drug: Loperamide
- Loperamide + Abemaciclib (Experimental): Cohort 2, only. 8 mg Loperamide co-administered with abemaciclib given orally once in up to 1 of 4 study periods.
  Interventions: Drug: Abemaciclib; Drug: Loperamide
- Loperamide + Placebo (Active Comparator): Cohort 2, only. 8 mg Loperamide co-administered with placebo given orally once in up to 1 of 4 study periods.
  Interventions: Drug: Placebo; Drug: Loperamide

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: Abemaciclib; Loperamide + Abemaciclib
Drug: Placebo — Administered orally
  Arms: Loperamide + Placebo; Placebo
Drug: Loperamide — Administered orally
  Arms: Loperamide; Loperamide + Abemaciclib; Loperamide + Placebo

SUMMARY:
The purposes of this study are to determine:

* The effect of single increasing doses of the study drug, abemaciclib, on healthy participants.
* The relationship between the amount of abemaciclib and the electrical tracing of the heart rhythm when abemaciclib is given.
* How much abemaciclib is found in the bloodstream and how long the body takes to get rid of it.

Information about any side effects that occur will be collected. The study will enroll two groups (cohorts) of participants. Each group will complete 4 study periods. This study is expected to last about 3 months. Screening may occur up to 28 days prior to enrollment. All participants will undergo a follow-up assessment approximately 21 days after administration of their final dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or females, as determined by medical history and physical examination

  * Male participants will be sterile
  * Female participants must not be of childbearing potential

Exclusion Criteria:

* Have known allergies to abemaciclib, related compounds, or any components of the formulation
* Have an abnormality in the 12-lead electrocardiogram (ECG) including a Fridericia's corrected QT interval (QTcF) greater than 450 milliseconds (ms) (males) or greater than 470 ms (females)
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs
* Have a gastrointestinal disorder causing clinically significant symptoms such as nausea, vomiting, and diarrhea, or malabsorption syndromes, or constipation

Additional Exclusion Criterion for Participants Enrolled in Cohort 2:

* Have a known hypersensitivity to loperamide hydrochloride or to any of the excipients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Covance Clinical Research Unit, Daytona Beach, Florida
  - Covance Clinical Research Unit, Evansville, Indiana

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dose escalation study with 2 cohorts, participants in cohort 1 were randomized to 1 of 4 sequences & participants in cohort 2 were randomized to 1 of 3 sequences. Cohort 1 had periods 1 to 4 with at least 5 days washout between each dose, Cohort 2 had periods 4(DDI) to 7 with at least 8 days washout between each dose.
Groups:
- Cohort 1 Sequence 1: Abemaciclib or matching placebo was administered orally on day 1 of each period based on below dosing schedule:
  Period 1- Placebo; Period 2- 200 milligram (mg) Abemaciclib; Period 3- 300 mg Abemaciclib; Period 4- 400 mg Abemaciclib.
- Cohort 1 Sequence 2: Abemaciclib or matching placebo was administered orally on day 1 of each period based on below dosing schedule:
  Period 1- 200 mg Abemaciclib; Period 2- Placebo; Period 3- 300 mg Abemaciclib; Period 4- 400 mg Abemaciclib.
- Cohort 1 Sequence 3: Abemaciclib matching placebo was administered orally on day 1 of each period based on below dosing schedule.
  Period 1- 200 mg Abemaciclib; Period 2- 300 mg Abemaciclib; Period 3- Placebo; Period 4- 400 mg Abemaciclib.
- Cohort 1 Sequence 4: Abemaciclib or matching placebo was administered orally on day 1 of each period based on below dosing schedule:
  Period 1- 200 mg Abemaciclib; Period 2- 300 mg Abemaciclib; Period 3- 400 mg Abemaciclib; Period 4- Placebo.
- Cohort 2 Sequence 1: Abemaciclib or matching placebo was administered orally on day 1 of each period based on below dosing schedule:
  Period 4 (DDI)- 8 mg Loperamide (on day -3 & 1) & Placebo; Period 5- Placebo; Period 6- 400 mg Abemaciclib; Period 7- 600 mg Abemaciclib.
- Cohort 2 Sequence 2: Abemaciclib or matching placebo was administered orally on day 1 of each period based on below dosing schedule:
  Period 4 (DDI)- 8 mg Loperamide (on Day -3 & 1) & 400 mg Abemaciclib; Period 5- 400 mg Abemaciclib; Period 6- Placebo; Period 7- 600 mg Abemaciclib.
- Cohort 2 Sequence 3: Abemaciclib or matching placebo was administered orally on day 1 of each period based on below dosing schedule:
  Period 4 (DDI)- 8 mg Loperamide (on day -3 & 1) & 400 mg Abemaciclib; Period 5- 400 mg Abemaciclib; Period 6- 600 mg Abemaciclib; Period 7- Placebo.
Period: Period 1
Arm/Group | Cohort 1 Sequence 1 | Cohort 1 Sequence 2 | Cohort 1 Sequence 3 | Cohort 1 Sequence 4 | Cohort 2 Sequence 1 | Cohort 2 Sequence 2 | Cohort 2 Sequence 3
Started | 5 | 5 | 5 | 5 | 0 | 0 | 0
Completed | 5 | 5 | 5 | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Cohort 1 Sequence 1 | Cohort 1 Sequence 2 | Cohort 1 Sequence 3 | Cohort 1 Sequence 4 | Cohort 2 Sequence 1 | Cohort 2 Sequence 2 | Cohort 2 Sequence 3
Started | 5 | 5 | 5 | 5 | 0 | 0 | 0
Completed | 5 | 5 | 5 | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Cohort 1 Sequence 1 | Cohort 1 Sequence 2 | Cohort 1 Sequence 3 | Cohort 1 Sequence 4 | Cohort 2 Sequence 1 | Cohort 2 Sequence 2 | Cohort 2 Sequence 3
Started | 5 | 5 | 5 | 5 | 0 | 0 | 0
Completed | 5 | 5 | 5 | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 4
Arm/Group | Cohort 1 Sequence 1 | Cohort 1 Sequence 2 | Cohort 1 Sequence 3 | Cohort 1 Sequence 4 | Cohort 2 Sequence 1 | Cohort 2 Sequence 2 | Cohort 2 Sequence 3
Started | 5 | 5 | 5 | 4 | 0 | 0 | 0
Completed | 5 | 5 | 5 | 4 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4 (DDI)
Arm/Group | Cohort 1 Sequence 1 | Cohort 1 Sequence 2 | Cohort 1 Sequence 3 | Cohort 1 Sequence 4 | Cohort 2 Sequence 1 | Cohort 2 Sequence 2 | Cohort 2 Sequence 3
Started (Participants were mutually exclusive of cohorts, Participants in Cohort 1 & 2 are different.) | 0 | 0 | 0 | 0 | 7 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 7 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Cohort 1 Sequence 1 | Cohort 1 Sequence 2 | Cohort 1 Sequence 3 | Cohort 1 Sequence 4 | Cohort 2 Sequence 1 | Cohort 2 Sequence 2 | Cohort 2 Sequence 3
Started | 0 | 0 | 0 | 0 | 7 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 7 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 6
Arm/Group | Cohort 1 Sequence 1 | Cohort 1 Sequence 2 | Cohort 1 Sequence 3 | Cohort 1 Sequence 4 | Cohort 2 Sequence 1 | Cohort 2 Sequence 2 | Cohort 2 Sequence 3
Started | 0 | 0 | 0 | 0 | 7 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 7 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 7
Arm/Group | Cohort 1 Sequence 1 | Cohort 1 Sequence 2 | Cohort 1 Sequence 3 | Cohort 1 Sequence 4 | Cohort 2 Sequence 1 | Cohort 2 Sequence 2 | Cohort 2 Sequence 3
Started | 0 | 0 | 0 | 0 | 7 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 7 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Single ascending doses of 200, 300, and 400 mg of Abemaciclib & Placebo were administered orally in one of the four sequences in each period.
- Cohort 2: Single ascending doses of 400, 600 mg Abemaciclib & Placebo were administered orally in one of the four sequences in each period. Loperamide 8mg was administered orally in period 4 (DDI) along with Abemaciclib.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 20 | 15 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (7.9) | 58 (7.5) | 52.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 18 | 14 | 32
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 15 | 35
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 0 | 10
  Not Hispanic or Latino | 10 | 15 | 25
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilogram per square meter (Kg/m^2)] | 26.80 (3.15) | 27.55 (2.35) | 27.12 (2.82)

OUTCOME MEASURES:

1. Primary Outcome: Mean Time Matched Placebo-Adjusted Changes From Baseline For Fridericia's Corrected QT Interval (ΔΔQTcF)
Description: QT interval is a measure of the time between the start of the Q wave and the end of the T wave and was calculated from electrocardiogram (ECG) data. ECG monitoring was conducted using a 12-lead digital Holter recorder from approximately 2 hours predose through 24 hours postdose on Day 1 of each period using 12-lead digital Holter recorder.
  Fridericia-corrected QT interval (QTcF): QTcF = QT/RR1/3, where RR is the interval between two R waves.
Time Frame: Day 1: 2hr,4hr,6hr,8hr,10hr,12hr,14hr,24hr Post Dose
Population: All randomized participants who received at least one dose of study drug and had baseline and post baseline QTcF values.
Measure: Mean (90% Confidence Interval); unit: Millisecond (msec)
Groups:
- 200 mg Abemaciclib: 200 mg Abemaciclib was given orally.
- 300 mg Abemaciclib: 300 mg Abemaciclib was given orally.
- 400 mg Abemaciclib: 400mg Abemaciclib was given orally.
- 600 mg Abemaciclib: 600 mg Abemaciclib was given orally.
Arm/Group | 200 mg Abemaciclib | 300 mg Abemaciclib | 400 mg Abemaciclib | 600 mg Abemaciclib
Number analyzed (Participants) | 19 | 19 | 33 | 15
Millisecond (msec)
  2hr: number analyzed (Participants) | 18 | 19 | 33 | 15
  2hr | 1.4 [-0.4 to 4.8] | 3.3 [-2.1 to 4.3] | 0.2 [-3.7 to 1.3] | -2.1 [-7.3 to 0.6]
  4hr: number analyzed (Participants) | 19 | 18 | 33 | 15
  4hr | -2.0 [-5.1 to 1.6] | 0.8 [-4.5 to 0.8] | -0.7 [-4.9 to 0.6] | -4.2 [-9.9 to 0.9]
  6hr: number analyzed (Participants) | 17 | 17 | 31 | 14
  6hr | 0.6 [-1.5 to 5.2] | -0.2 [-5.8 to 1.2] | -1.8 [-5.9 to -0.1] | -3.7 [-10.3 to -0.8]
  8hr: number analyzed (Participants) | 18 | 19 | 31 | 14
  8hr | 2.8 [0.7 to 6.4] | 2.7 [-3.1 to 4.0] | 2.2 [-1.8 to 3.5] | 2.8 [-3.9 to 5.8]
  10hr: number analyzed (Participants) | 18 | 19 | 31 | 14
  10hr | 2.1 [0.6 to 5.1] | 1.3 [-3.7 to 1.7] | 1.5 [-2.4 to 2.1] | 5.9 [-2.8 to 11]
  12hr: number analyzed (Participants) | 18 | 19 | 32 | 15
  12hr | -0.3 [-4.7 to 5.6] | -0.7 [-6.6 to 0.8] | -0.5 [-4.4 to 0.1] | 4.4 [-0.9 to 7.2]
  14hr: number analyzed (Participants) | 18 | 19 | 31 | 14
  14hr | 3.9 [1.4 to 7.9] | 3.3 [-2.1 to 4.1] | 1.0 [-3.9 to 2.6] | 2.3 [-4.4 to 5.4]
  24hr: number analyzed (Participants) | 18 | 18 | 31 | 14
  24hr | 1.4 [-1.2 to 5.5] | 4.2 [-0.7 to 4.8] | -0.4 [-4.7 to 1.3] | 0.9 [-7.1 to 4.6]

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Abemaciclib
Description: Blood samples were collected from participants in Cohort 1(all periods) and Cohort 2 (Periods 5, 6, and 7) to determine the plasma concentrations of Abemaciclib.
Time Frame: Day 1: 2, 4, 6, 8, 10, 12, 14, 24, 48, 72, 96, and 120 hours Post Dose
Population: All randomized participants who received at least one dose of study drug in Cohort 1 all periods & Cohort 2 periods 5,6, and 7 with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per Milliliter (ng/mL)
Groups:
- 400 mg Abemaciclib: 400 mg Abemaciclib was given orally.
- 400 mg Abemaciclib + Loperamide 8mg: 400 mg Abemaciclib was given orally along with 8mg Loperamide.
Arm/Group | 200 mg Abemaciclib | 300 mg Abemaciclib | 400 mg Abemaciclib | 600 mg Abemaciclib | 400 mg Abemaciclib + Loperamide 8mg
Number analyzed (Participants) | 19 | 20 | 31 | 8 | 7
Nanogram per Milliliter (ng/mL) | 102 (31) | 130 (40) | 182 (42) | 308 (45) | 199 (55)

3. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time 0 to Last Time Point With Measurable Concentration AUC(0-tlast) of Abemaciclib
Description: Blood samples were collected from participants in Cohort 1(all periods) and Cohort 2 (Periods 5, 6, and 7) to determine the plasma concentrations of Abemaciclib 0-tlast.
Time Frame: Day 1: 2, 4, 6, 8, 10, 12, 14, 24, 48, 72, 96, and 120 hours Post Dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- 400 mg Abemaciclib + 8 mg Loperamide: 400 mg Abemaciclib was given orally along with 8 mg Loperamide.
Arm/Group | 200 mg Abemaciclib | 300 mg Abemaciclib | 400 mg Abemaciclib | 600 mg Abemaciclib | 400 mg Abemaciclib + 8 mg Loperamide
Number analyzed (Participants) | 19 | 20 | 31 | 8 | 7
ng*hr/mL | 3560 (38) | 5210 (37) | 7610 (46) | 14600 (42) | 9420 (57)

4. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Last Time Point With Measurable Concentration [AUC(0-tlast)] of Loperamide
Description: Blood samples were collected from participants in Cohort 2 Period 4 (DDI) to determine plasma concentrations of Loperamide.
Time Frame: Day -3: Predose, 1, 2, 4, 6, 8, 12, 14, 24, and 48 hours postdose;Day 1 predose, (-0.25 hours), and Day1: 1, 2, 4, 6, 8, 10, 12, 14, 24, 48, and 72 hours Post Dose
Population: All randomized participants in Cohort 2 Period 4 (DDI) who received Loperamide & had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Groups:
- 8 mg Loperamide: 8 mg Loperamide was given orally.
- 8 mg Loperamide + 400 mg Abemaciclib: 8 mg Loperamide was given orally along with 400 mg Abemaciclib.
Arm/Group | 8 mg Loperamide | 8 mg Loperamide + 400 mg Abemaciclib
Number analyzed (Participants) | 18 | 7
ng*hr/mL | 46.1 (47) | 47.3 (53)

5. Secondary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Loperamide
Description: as for outcome 4
Time Frame: Day -3: Predose,1, 2, 4, 6, 8, 12, 14, 24, and 48 hours postdose;Day 1 predose, (-0.25 hours), and Day1: 1, 2, 4, 6, 8, 10, 12, 14, 24, 48, and 72 hours Post Dose
Population: All randomized participants in Cohort 2 Period 4 (DDI) who received Loperamide & had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 8 mg Loperamide | 8 mg Loperamide + 400 mg Abemaciclib
Number analyzed (Participants) | 18 | 7
ng/mL | 1.83 (56) | 2.17 (49)

ADVERSE EVENTS:
Time Frame: Up to 117 days
Description: All randomized participants who received at least once dose study drug.
Groups:
- Placebo: Matching placebo was given orally in place of Abemaciclib.
- 8 mg Loperamide + Placebo: 8 mg Loperamide was given orally & matching placebo was used for Abemaciclib
- 8 mg Loperamide + 400 mg Abemaciclib: 400 mg Abemaciclib was given orally along with 8 mg Loperamide.
Arm/Group | Placebo | 200 mg Abemaciclib | 300 mg Abemaciclib | 400 mg Abemaciclib | 600 mg Abemaciclib | 8 mg Loperamide | 8 mg Loperamide + Placebo | 8 mg Loperamide + 400 mg Abemaciclib
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/20 | 0/20 | 0/35 | 0/15 | 0/15 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 9/34 | 4/20 | 5/20 | 17/35 | 12/15 | 5/15 | 3/7 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=34) | 200 mg Abemaciclib (N=20) | 300 mg Abemaciclib (N=20) | 400 mg Abemaciclib (N=35) | 600 mg Abemaciclib (N=15) | 8 mg Loperamide (N=15) | 8 mg Loperamide + Placebo (N=7) | 8 mg Loperamide + 400 mg Abemaciclib (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 4 (4) | 11 (11) | 11 (13) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 6 (6) | 8 (9) | 0 (0) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 1 (1)
Application site irritation (General disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenderness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
At the 600-mg dose level, the protocol-specified dose escalation stopping criteria had been met so no participants received the 900-mg dose in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days